CLINICAL TRIAL: NCT00099411
Title: Myocardial Viability and Remodeling in the Occluded Artery Trial (OAT)-Ancillary to OAT
Brief Title: Heart Muscle Viability and Remodeling in Individuals Post-Heart Attack
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1279; R01HL075456 (NIH)
Record Dates: First submitted 2004-12-13; First posted 2004-12-14 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases; Heart Failure, Congestive
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the effect of heart muscle viability on left ventricular (LV) remodeling after a heart attack; to explore the relationships between retained viability of the area of tissue death (infarct zone), LV remodeling, response to the Occluded Artery Trial (OAT) intervention, and response to late percutaneous coronary intervention of the infarct related artery (IRA).

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease is a major health problem in the United States. It is estimated that in 2003, more than 600,000 Americans had a new heart attack, and more than 400,000 experienced a recurrent heart attack. Up to 40% of individuals with a new or recurrent heart attack will show a complete occlusion, or blocking, of the IRA on follow-up angiography. Many people with an occluded IRA post-heart attack are at risk for progressive LV remodeling in the heart, which can lead to congestive heart failure.

The NHLBI-funded OAT study is testing the hypothesis that opening an occluded IRA 3 to 28 days following a heart attack will reduce the composite endpoint of mortality, recurrent heart attack, and New York Heart Association class IV heart failure over a three-year follow-up period. OAT has enrolled approximately 1,100 participants at 240 centers in 24 countries. Among the mechanisms proposed to explain the benefit of late revascularization, recovery of LV function and attenuation of LV remodeling due to restoration of blood flow to viable myocardium, or heart muscle, is the most plausible.

DESIGN NARRATIVE:

An estimated 200 individuals who have had a heart attack will be enrolled in this study. The primary aims of this study are the following: 1) to test the hypothesis that participants who demonstrate preservation of viability within the infarct zone will have less progressive remodeling compared to participants exhibiting predominant infarct, and 2) to test the hypothesis that preservation of viability will modify the treatment effect of randomization to late revascularization in participants with an occluded IRA 3 to 28 days after the heart attack. All participants will have resting gated Tc-99m sestamibi SPECT imaging at baseline, and again 1 year later. Parameters of baseline viability within the infarct zone, and serial measures of LV volume change and function will be centrally assessed by the Cardiac Imaging Core Laboratory at Tufts Medical Center. The major study endpoint to address the hypotheses will be serial change in LV end-diastolic volume, based on the degree of preservation of viability within the defined infarct zone. Sample size calculations will be based on data evaluated by the same group from a similar number of participants studied at a similar number of clinical sites.

ELIGIBILITY:
Inclusion Criteria:

* Has experienced a heart attack 3 to 28 days prior to study entry
* Has an occluded IRA at catheterization

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who have experienced a heart attack 3 to 28 days prior to study entry.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2007-06-30 (Actual); Study Completion 2007-06-30 (Actual)

PRIMARY OUTCOMES:
The primary end point of LV remodeling was assessed by change in LV EDV from baseline to 1 year. | 1 year
  The primary end point of LV remodeling was assessed by change in LV EDV from baseline to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: James E. Udelson, Study Chair — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No